CLINICAL TRIAL: NCT04277650
Title: System for High Intensity EvaLuation During Radiation Therapy (SHIELD-RT): A Prospective Randomized Study of Machine Learning-directed Clinical Evaluations During Outpatient Cancer Radiation and Chemoradiation
Brief Title: System for High-Intensity Evaluation During Radiotherapy
Acronym: SHIELD-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00100647
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-01

CONDITIONS: Radiation Therapy Complication; Chemotherapeutic Toxicity
MeSH Terms: interventions — Machine Learning Algorithms

STUDY DESIGN:
Intervention Model Description: Participants identified by the machine learning (ML) algorithm as high risk were randomized to either once weekly or twice weekly clinical evaluations
Masking Description: The ML directed twice-weekly evaluation arm was unblinded. Participants and providers were blinded to ML identification of high risk participants in the once weekly evaluation (standard of care) arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once weekly clinical evaluation (Active Comparator): Outpatient participants evaluated as high risk by the machine learning algorithm and provided once weekly clinical evaluations
  Interventions: Other: Machine learning algorithm
- Twice weekly clinical evaluation (Experimental): Outpatient participants evaluated as high risk by the machine learning algorithm and provided twice weekly clinical evaluations
  Interventions: Other: Machine learning algorithm

INTERVENTIONS:
Other: Machine learning algorithm — machine learning directed identification of radiotherapy or chemoradiotherapy patients at high-risk for emergency department acute care and/or hospitalization

SUMMARY:
This quality improvement project will evaluate the implementation of a previously described intervention (twice per week on-treatment clinical evaluations) in a feasible fashion using a previously described machine learning algorithm identifying patients identified at high risk for an emergency visit or hospitalization during radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

• started outpatient radiation therapy with or without concurrent systemic therapy at Duke Cancer Center

Exclusion Criteria:

* undergoing total body radiation therapy for hematopoetic stem cell transplantation
* undergoing therapy as inpatient
* treating physician who opted out of randomization
* completed radiation therapy prior to algorithm execution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of unplanned emergency department visits or hospital admissions | 6 months

SECONDARY OUTCOMES:
Number of unplanned emergency department visits or hospital admissions up to 15 days post radiation treatment | up to 15 days post radiation treatment
Number of missed clinical evaluation visits | 6 months
Number of acute care visits with listed reason as anemia, nutrition (including dehydration), diarrhea, emesis, infectious (including fever, pneumonia, and sepsis), nausea, neutropenia, pain category | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified summary data in the form of publication data tables and figures will be shared. Individual level data will not be shared.

REFERENCES:
- [Result] Hong JC, Eclov NCW, Dalal NH, Thomas SM, Stephens SJ, Malicki M, Shields S, Cobb A, Mowery YM, Niedzwiecki D, Tenenbaum JD, Palta M. System for High-Intensity Evaluation During Radiation Therapy (SHIELD-RT): A Prospective Randomized Study of Machine Learning-Directed Clinical Evaluations During Radiation and Chemoradiation. J Clin Oncol. 2020 Nov 1;38(31):3652-3661. doi: 10.1200/JCO.20.01688. Epub 2020 Sep 4. PMID 32886536
- [Derived] James B Yu Md Mhs Fastro, Hong JC. AI Use in Prostate Cancer: Potential Improvements in Treatments and Patient Care. Oncology (Williston Park). 2024 May 13;38(5):208-209. doi: 10.46883/2024.25921021. PMID 38776517
- [Derived] Natesan D, Eisenstein EL, Thomas SM, Eclov NCW, Dalal NH, Stephens SJ, Malicki M, Shields S, Cobb A, Mowery YM, Niedzwiecki D, Tenenbaum JD, Palta M, Hong JC. Health Care Cost Reductions with Machine Learning-Directed Evaluations during Radiation Therapy - An Economic Analysis of a Randomized Controlled Study. NEJM AI. 2024 Apr;1(4):10.1056/aioa2300118. doi: 10.1056/aioa2300118. Epub 2024 Mar 15. PMID 38586278
- [Derived] Hong JC, Eclov NCW, Stephens SJ, Mowery YM, Palta M. Implementation of machine learning in the clinic: challenges and lessons in prospective deployment from the System for High Intensity EvaLuation During Radiation Therapy (SHIELD-RT) randomized controlled study. BMC Bioinformatics. 2022 Sep 30;23(Suppl 12):408. doi: 10.1186/s12859-022-04940-3. PMID 36180836